CLINICAL TRIAL: NCT04068896
Title: A Phase 1/2 Dose-Finding Study Followed by Expansion Cohorts of NGM120, a GFRAL Antagonist Monoclonal Antibody Blocking GDF15 Signaling, in Subjects With Advanced Solid Tumors and Pancreatic Cancer Using Combination Therapy
Brief Title: Study of NGM120 in Subjects With Advanced Solid Tumors, Pancreatic Cancer, and Prostate Cancer Using Combination Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-0402
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cancer; Metastatic Castration-resistant Prostate Cancer; Bladder Cancer; Melanoma; Non-small Cell Lung Cancer; Colorectal Cancer; Gastric Cancer; Esophageal Cancer; Ovarian Cancer; Head Neck Squamous Cell Carcinoma; Prostate Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Urinary Bladder Neoplasms; Melanoma; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Ovarian Neoplasms; Squamous Cell Carcinoma of Head and Neck; Prostatic Neoplasms | interventions — Gemcitabine; Albumin-Bound Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1 NGM120 30mg (Experimental): NGM120 30mg Subcutaneous Injection
  Interventions: Biological: NGM120 30mg
- Part 1 NGM120 100mg (Experimental): NGM120 100mg Subcutaneous Injection
  Interventions: Biological: NGM120 100mg
- Part 2 NGM120 30mg (Experimental): NGM120 30mg Subcutaneous Injection together with gemcitabine (1000 mg/m2 weekly for first 3 weeks of the 4-week cycle) and Abraxane (125 mg/m2 weekly for first 3 weeks of the 4-week cycle).
  Interventions: Biological: NGM120 30mg with Gemcitabine and Abraxane
- Part 2 NGM120 100mg (Experimental): NGM120 100mg Subcutaneous Injection together with gemcitabine (1000 mg/m2 weekly for first 3 weeks of the 4-week cycle) and Abraxane (125 mg/m2 weekly for first 3 weeks of the 4-week cycle).
  Interventions: Biological: NGM120 100mg with Gemcitabine and Abraxane
- Part 3 NGM120 100mg Q3W (Experimental): NGM120 100mg Subcutaneous Injection NGM120 100mg Subcutaneous Injection every 3 weeks
  Interventions: Biological: NGM120 100mg Q3W
- Part 2 Placebo (Placebo Comparator): Placebo together with gemcitabine (1000 mg/m2 weekly for first 3 weeks of the 4-week cycle) and Abraxane (125 mg/m2 weekly for first 3 weeks of the 4-week cycle).
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: NGM120 30mg — NGM120 30mg Subcutaneous Injection
  Arms: Part 1 NGM120 30mg
Biological: NGM120 100mg — NGM120 100mg Subcutaneous Injection
  Arms: Part 1 NGM120 100mg
Biological: NGM120 30mg with Gemcitabine and Abraxane — NGM120 30mg Subcutaneous Injection together with gemcitabine (1000 mg/m2 weekly for first 3 weeks of the 4-week cycle) and Abraxane (125 mg/m2 weekly for first 3 weeks of the 4-week cycle).
  Arms: Part 2 NGM120 30mg
Biological: NGM120 100mg with Gemcitabine and Abraxane — NGM120 100 mg Subcutaneous Injection together with gemcitabine (1000 mg/m2 weekly for first 3 weeks of the 4-week cycle) and Abraxane (125 mg/m2 weekly for first 3 weeks of the 4-week cycle).
  Arms: Part 2 NGM120 100mg
Biological: NGM120 100mg Q3W — NGM120 100mg Subcutaneous Injection every 3 weeks
  Arms: Part 3 NGM120 100mg Q3W
Other: Placebo — Placebo
  Arms: Part 2 Placebo

SUMMARY:
Study of NGM120 in subjects with advanced solid tumors and pancreatic cancer (Part 1 and 2) and metastatic castration resistant prostate cancer (Part 3).

DETAILED DESCRIPTION:
The aim of the study is to evaluate the safety and tolerability of NGM120 monotherapy in subjects with select advanced solid tumors (Part 1), NGM120 in combination with gemcitabine and Abraxane for the management of metastatic pancreatic cancer (Part 2), and NGM120 in metastatic castration-resistant prostate cancer (mCRPC) patients who have progressed under 1 or more lines of ADT (Part 3), for up to 24 months of treatment.

ELIGIBILITY:
Inclusion Criteria (Part 1 and 2):

1. Have histologically confirmed metastatic pancreatic adenocarcinoma. Recurrent unresectable pancreatic cancer is acceptable as long as the treatment is first-line.
2. Have not received any approved chemotherapy, except in the adjuvant setting.
3. Life expectancy of at least 12 weeks
4. Male subjects must agree to use contraception as per protocol during the treatment period and for at least 90 days after the last study treatment administration and refrain from donating sperm during this period.
5. Provision of an archival tumor sample (within 5 years). If an archival sample is unavailable, a fresh biopsy can be obtained during Screening. If archival tissue or biopsy sample is unavailable, the subject is ineligible.

Inclusion Criteria (Part 3 Prostate Cancer):

1. Metastatic, castrate resistance, histologically confirmed prostate cancer; continuous medical castration for ≥8 weeks prior to screening.
2. Effective castration with serum testosterone levels <0.5 ng/mL (50 ng/dL; 1.7 nmol/L).
3. Have serum GDF15 levels ≥1300 pg/mL.
4. Have experienced PSA progression under 1 or more lines of ADT in the absence or presence of radiographic and/or clinical progression, who decline or are not eligible to receive chemotherapy.
5. Have had PSA doubling time of >3 months.

Exclusion Criteria (All parts):

1. Subject was using immunosuppressive medications within 14 days before Screening with the exception of topical (intranasal, inhaled, and local injection), systemic (prednisone equivalent 10 mg/day or less), or as needed for hypersensitivity reactions such as computed tomography (CT) scan premedication.
2. Subject has active infections or other serious underlying significant medical illness, abnormal and clinically significant laboratory findings or psychiatric illness/social situation.
3. Subject is using a pacemaker, implantable cardiac defibrillator, neurostimulator, cochlear implants, cochlear implants, or other electronic medical equipment.
4. Subject has documented immunodeficiency or organ transplant.
5. Subject has an untreated central nervous system disease, leptomeningeal disease or cord compression.
6. Subject has a history, or presence, of significant cardiovascular diseases; including uncontrolled hypertension, clinically relevant cardiac arrhythmia, unstable angina or myocardial infarction within 6 months before randomization, congestive heart failure > New York Heart Association Class II, severe peripheral vascular disease, corrected QT (QTc) prolongation >470 msec, clinically significant pericardial effusion.
7. Subject has a history or presence of documented inflammatory bowel disease.
8. Subject is known to be positive for human immunodeficiency virus (HIV) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2024-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NGM Study Director, Study Director — NGM Biopharmaceuticals, Inc
Locations (19):
- United States (19):
  - NGM Clinical Study Site, Tucson, Arizona
  - NGM Clinical Study Site, Los Angeles, California
  - NGM Clinical Study Site, Sacramento, California
  - NGM Clinical Study Site, San Diego, California
  - NGM Clinical Study Site, Santa Monica, California
  - NGM Clinical Study Site, Aurora, Colorado
  - NGM Clinical Study Site, Washington D.C., District of Columbia
  - NGM Clinical Study Site, Miami, Florida
  - NGM Clinical Study Site, Chicago, Illinois
  - NGM Clinical Study Site, Baltimore, Maryland
  - NGM Clinical Study Site, Cincinnati, Ohio
  - NGM Clinical Study Site, Philadelphia, Pennsylvania
  - NGM Clinical Study Site, Charleston, South Carolina
  - NGM Clinical Study Site, Myrtle Beach, South Carolina
  - NGM Clinical Study Site, Nashville, Tennessee
  - NGM Clinical Study Site, Dallas, Texas
  - NGM Clinical Study Site, Houston, Texas
  - NGM Clinical Study Site, Seattle, Washington
  - NGM Clinical Study Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 89 patients were enrolled (signed consent), however only 87 patients received at least 1 dose of study treatment. The participant flow contains information from these 87 treated patients, that are also considered the Safety Analysis set for CSR and study results
Groups:
- Part 1 NGM120 30 mg: NGM120 30 mg Subcutaneous Injection
- Part 1 NGM120 100 mg; Part 3 NGM120 100 mg: NGM120 100 mg Subcutaneous Injection
- Part 2 NGM120 30 mg: NGM120 30 mg Subcutaneous Injection together with gemcitabine (1000 mg/m2 weekly for first 3 weeks of the 4-week cycle) and Abraxane (125 mg/m2 weekly for first 3 weeks of the 4-week cycle).
- Part 2 NGM120 100 mg: NGM120 100 mg Subcutaneous Injection together with gemcitabine (1000 mg/m2 weekly for first 3 weeks of the 4-week cycle) and Abraxane (125 mg/m2 weekly for first 3 weeks of the 4-week cycle).
- Part 2 Placebo: Placebo subcutaneous injection together with gemcitabine (1000 mg/m2 weekly for first 3 weeks of the 4-week cycle) and Abraxane (125 mg/m2 weekly for first 3 weeks of the 4-week cycle).
Period: Overall Study
Arm/Group | Part 1 NGM120 30 mg | Part 1 NGM120 100 mg | Part 2 NGM120 30 mg | Part 2 NGM120 100 mg | Part 2 Placebo | Part 3 NGM120 100 mg
Started | 10 | 10 | 10 | 31 | 20 | 6
Completed | 0 | 1 | 2 | 4 | 0 | 0
Not Completed | 10 | 9 | 8 | 27 | 20 | 6
Not completed — Adverse Event | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 3 | 1 | 3 | 19 | 17 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0
Not completed — progressive disease | 3 | 5 | 3 | 2 | 1 | 2
Not completed — Study terminated by sponsor | 0 | 0 | 1 | 2 | 1 | 4
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 2 | 1 | 0
Not completed — Symptomatic deterioration | 2 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1 NGM120 100mg; Part 3 NGM120 100mg: NGM120 100 mg Subcutaneous Injection
- Part 2 NGM120 100mg: NGM120 100 mg Subcutaneous Injection together with gemcitabine (1000 mg/m2 weekly for first 3 weeks of the 4-week cycle) and Abraxane (125 mg/m2 weekly for first 3 weeks of the 4-week cycle).
- Total: Total of all reporting groups
Arm/Group | Part 1 NGM120 30mg | Part 1 NGM120 100mg | Part 2 NGM120 30mg | Part 2 NGM120 100mg | Part 2 Placebo | Part 3 NGM120 100mg | Total
Number analyzed (Participants) | 10 | 10 | 10 | 31 | 20 | 6 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 2 | 2 | 11 | 4 | 1 | 27
  >=65 years | 3 | 8 | 8 | 20 | 16 | 5 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (9.08) | 65.6 (12.21) | 67.7 (8.27) | 67.0 (9.06) | 69.9 (8.10) | 69.0 (11.92) | 67.2 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 8 | 13 | 11 | 0 | 37
  Male | 6 | 9 | 2 | 18 | 9 | 6 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 2 | 0 | 1 | 1 | 7
  Not Hispanic or Latino | 8 | 9 | 7 | 30 | 15 | 4 | 73
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 4 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 2 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 2 | 0 | 3
  Black or African American | 0 | 2 | 1 | 4 | 0 | 1 | 8
  White | 8 | 8 | 4 | 17 | 11 | 5 | 53
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 5 | 7 | 6 | 0 | 19
BMI [Mean (Standard Deviation); unit: kg/m2] | 24.93 (5.759) | 26.46 (4.636) | 26.53 (9.694) | 25.72 (5.119) | 25.04 (5.113) | 31.20 (5.852) | 26.03 (5.89)
Metastatic Disease [Count of Participants; unit: Participants]
  Yes | 9 | 10 | 10 | 29 | 19 | 6 | 83
  No | 1 | 0 | 0 | 2 | 1 | 0 | 4
Sites of Metastases [Number; unit: count of metastatic sites]
  Bone | 3 | 6 | 1 | 1 | 0 | 5 | 16
  Liver | 5 | 4 | 5 | 17 | 16 | 0 | 47
  Lung | 2 | 4 | 4 | 10 | 5 | 1 | 26
  Peritoneum | 2 | 0 | 2 | 2 | 0 | 0 | 6
  Other | 2 | 2 | 1 | 5 | 3 | 2 | 15
Time from Initial cancer diagnosis [Mean (Standard Deviation); unit: Months] | 40.775 (21.0265) | 61.841 (67.6111) | 6.328 (12.9190) | 4.769 (7.4036) | 4.350 (6.1938) | 140.167 (69.4910) | 24.86 (47.45)

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Safety and Tolerability of NGM120 in Subjects
Description: Number of Participants with NGM120/Placebo-Related Treatment Emergent Adverse Events
Time Frame: From enrollment to end of treatment up to 24 months
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Groups:
- Part 3 NGM120 100mg: NGM120 100mg Subcutaneous Injection
Arm/Group | Part 1 NGM120 30mg | Part 1 NGM120 100mg | Part 2 NGM120 30mg | Part 2 NGM120 100mg | Part 2 Placebo | Part 3 NGM120 100mg
Number analyzed (Participants) | 10 | 10 | 10 | 31 | 20 | 6
Participants | 1 | 6 | 6 | 17 | 12 | 2

2. Primary Outcome: To Determine the Safety and Tolerability of NGM120
Description: Discontinuation of investigational product due to toxicity
Time Frame: From enrollment to end of treatment up to 24 months
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 NGM120 30mg | Part 1 NGM120 100mg | Part 2 NGM120 30mg | Part 2 NGM120 100mg | Part 2 Placebo | Part 3 NGM120 100mg
Number analyzed (Participants) | 10 | 10 | 10 | 31 | 20 | 6
Participants | 2 | 0 | 2 | 8 | 3 | 0

3. Primary Outcome: To Determine the Safety and Tolerability of NGM120
Description: Local injection-site symptom assessment as evidenced by incidence of injection-site reactions
Time Frame: From enrollment to end of treatment up to 24 months
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 NGM120 30mg | Part 1 NGM120 100mg | Part 2 NGM120 30mg | Part 2 NGM120 100mg | Part 2 Placebo | Part 3 NGM120 100mg
Number analyzed (Participants) | 10 | 10 | 10 | 31 | 20 | 6
Participants | 0 | 1 | 0 | 4 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years, 8 months.
Arm/Group | Part 1 NGM120 30mg | Part 1 NGM120 100mg | Part 2 NGM120 30mg | Part 2 NGM120 100mg | Part 2 Placebo | Part 3 NGM120 100mg
All-Cause Mortality (participants affected / at risk) | 3/10 | 1/10 | 3/10 | 19/31 | 17/20 | 0/6
Serious Adverse Events (participants affected / at risk) | 5/10 | 3/10 | 5/10 | 26/31 | 10/20 | 1/6
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 10/10 | 31/31 | 20/20 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 NGM120 30mg (N=10) | Part 1 NGM120 100mg (N=10) | Part 2 NGM120 30mg (N=10) | Part 2 NGM120 100mg (N=31) | Part 2 Placebo (N=20) | Part 3 NGM120 100mg (N=6)
Sepsis (Infections and infestations) | 2 | 1 | 1 | 3 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0
Skin Infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Prostatic Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Corona Virus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Obstruction Gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 3 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 (0) | 0 | 1 | 0 | 0 (0)
Radiation injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 (0) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Device occlusion (Product Issues) | 0 | 0 | 0 | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 NGM120 30mg (N=10) | Part 1 NGM120 100mg (N=10) | Part 2 NGM120 30mg (N=10) | Part 2 NGM120 100mg (N=31) | Part 2 Placebo (N=20) | Part 3 NGM120 100mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 5 | 16 | 11 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1 | 1 | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 7 | 6 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 4 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 2 | 9 | 4 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 7 | 15 | 8 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 4 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 7 | 13 | 8 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Steatorrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 3 | 5 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 4 | 5 | 4 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 4 | 5 | 4 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 4 | 3 | 2 | 0
Generalised oedema (General disorders) | 0 | 0 | 1 | 1 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 3 | 1 | 0 | 1
Injection site erythema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Injection site laceration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 1 | 3 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 2 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 4 | 0 | 1
Oedema peripheral (General disorders) | 2 | 2 | 7 | 13 | 7 | 2
Pain (General disorders) | 0 | 0 | 0 | 2 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 3 | 6 | 14 | 4 | 0
Fatigue (General disorders) | 4 | 2 | 7 | 22 | 11 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 4 | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 3 | 3 | 2 | 0
Amylase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 3 | 6 | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 1 | 4 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 3 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 4 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 4 | 0 | 1 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 1 | 1 | 5 | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 5 | 13 | 9 | 0
Platelet count decreased (Investigations) | 1 | 0 | 3 | 10 | 9 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 2 | 0 | 0
Weight decreased (Investigations) | 2 | 1 | 5 | 10 | 6 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 2 | 6 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 4 | 6 | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 6 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 5 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 4 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3 | 1 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 1 | 6 | 4 | 0
Headache (Nervous system disorders) | 1 | 2 | 5 | 6 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 5 | 9 | 6 | 0
Insomnia (Psychiatric disorders) | 3 | 2 | 0 | 4 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 2 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 12 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 6 | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 8 | 6 | 6 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 5 | 5 | 7 | 2
Hypotension (Vascular disorders) | 1 | 0 | 2 | 5 | 3 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 3 | 3 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 3 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 2 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 2 | 0 | 2 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 5 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 4 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 4 | 3 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 10 | 4 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 2 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 4 | 1 | 0
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 6 | 2 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 1 | 4 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 4 | 2 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 2 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 3 | 2 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 3 | 2 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 3 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 1 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 2 | 4 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Seasonal Allergy (Immune system disorders) | 0 | 0 | 0 | 2 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/96/NCT04068896/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT04068896/SAP_001.pdf